CLINICAL TRIAL: NCT00394953
Title: A Randomized, Controlled, Open Label, Multicenter, Parallel-group Study to Compare the Effect of Mircera With That of Darbepoetin Alfa, Administered Intravenously at Extended Dosing Intervals, for the Maintenance Treatment of Anemia in Patients With Chronic Kidney Disease Who Are on Hemodialysis
Brief Title: A Study of Mircera for the Maintenance Treatment of Anemia in Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH17847
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa; continuous erythropoietin receptor activator

ARMS (2):
- MIRCERA (Experimental): Eligible participants with anemia in CKD who were on hemodialysis will receive methoxy polyethylene glycol-epoetin beta (MIRCERA [RO0503821]) IV once every month up to 52 weeks. The starting dose of MIRCERA which will be administered during the treatment period will depend on the dose of darbepoetin alfa administered during screening period i.e., 120, 200 and 360 mcg for weekly darbepoetin alfa doses of <40, 40-80, and >80 mcg, respectively.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Darbepoetin Alfa (Active Comparator): Eligible participants with anemia in CKD who were on hemodialysis will receive darbepoetin alfa (Aranesp) IV once every two weeks up to 26 weeks and darbepoetin alfa IV twice the dose than earlier, once every month from Week 27 up to Week 52.
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — As prescribed, iv.
  Other Names: Aranesp
  Arms: Darbepoetin Alfa
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 120, 200 or 360 micrograms iv / month, starting dose
  Arms: MIRCERA

SUMMARY:
This 2 arm study will compare the efficacy and safety of Mircera and darbepoetin alfa, administered at extended dosing intervals, in the maintenance treatment of anemia in patients with chronic kidney disease (CKD) who are on hemodialysis. Eligible patients receiving once-weekly intravenous (IV) darbepoetin alfa maintenance treatment will be randomized to receive either intravenous Mircera once a month (at a starting dose of 120, 200 or 360 micrograms/month, depending on the weekly dose of darbepoetin alfa prior to start of study) or intravenous darbepoetin alfa every 2 weeks before switching to once monthly administration. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic renal anemia;
* hemodialysis 3 times weekly for >=12 weeks before screening, and during screening/baseline period;
* receiving darbepoetin alfa maintenance therapy for >=8 weeks before screening, and during screening/baseline period.

Exclusion Criteria:

* overt gastrointestinal bleeding within 8 weeks before screening or during screening/baseline period;
* transfusion of red blood cells within 8 weeks before screening or during screening/baseline period;
* active malignancy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (78):
- Australia (5):
  - Adelaide
  - Clayton
  - Gosford
  - Parkville
  - Woolloongabba
- Austria (2):
  - Linz
  - Vienna
- Belgium (3):
  - Aalst
  - Brussels
  - Roeselare
- Canada (8):
  - Calgary, Alberta
  - Hamilton, Ontario
  - Kitchener, Ontario
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Trois-Rivières, Quebec
- Denmark (3):
  - Aalborg
  - Hillerød
  - Roskilde
- Finland (2):
  - Tampere
  - Turku
- France (20):
  - Auch
  - Bordeaux
  - Boulogne
  - Castelnau-le-Lez
  - Cergy-Pontoise
  - Chamalières
  - Dijon
  - Fleury-Mérogis
  - Hérouville-Saint-Clair
  - La Tronche
  - Lyon
  - Montpellier
  - Nîmes
  - Paris
  - Reims
  - Rennes
  - Saint-Brieuc
  - Saint-Herblain
  - Saint-Ouen
  - Villeurbanne
- Germany (6):
  - Bad Hersfeld
  - Bonn
  - Dortmund
  - München
  - Stuttgart
  - Villingen-Schwenningen
- Italy (8):
  - Bologna
  - Como
  - Genova
  - Lecco
  - Modena
  - Pavia
  - Prato
  - Venezia
- Netherlands (2):
  - Amsterdam
  - Dordrecht
- Leiria, Portugal
- Spain (10):
  - Alicante
  - Badalona
  - Barcelona
  - Bilbao
  - Córdoba
  - León
  - Madrid
  - Ourense
  - Santander
  - Vigo
- Switzerland (2):
  - Aarau
  - Lausanne
- United Kingdom (6):
  - Belfast
  - Canterbury
  - Glasgow
  - London
  - Manchester
  - Truro

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Carrera F, Lok CE, de Francisco A, Locatelli F, Mann JF, Canaud B, Kerr PG, Macdougall IC, Besarab A, Villa G, Kazes I, Van Vlem B, Jolly S, Beyer U, Dougherty FC; PATRONUS Investigators. Maintenance treatment of renal anaemia in haemodialysis patients with methoxy polyethylene glycol-epoetin beta versus darbepoetin alfa administered monthly: a randomized comparative trial. Nephrol Dial Transplant. 2010 Dec;25(12):4009-17. doi: 10.1093/ndt/gfq305. Epub 2010 Jun 3. PMID 20522670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 20 December 2006 to 27 November 2008 in Europe along with Canada and Australia. A total of 490 eligible participants were enrolled.
Pre-assignment Details: Out of 490 participants, one did not receive the study drug and was excluded from the safety population.
Groups:
- MIRCERA: Participants with anemia in chronic kidney disease (CKD) who were on hemodialysis received methoxy polyethylene glycol-epoetin beta (MIRCERA [RO0503821]) intravenously (IV) once every month up to 52 weeks. The starting dose of MIRCERA administered during the treatment period was dependent on the dose of darbepoetin alfa administered during screening period and was 120, 200 and 360 microgram per month (mcg/month) for weekly darbepoetin alfa doses of <40, 40-80, and >80 mcg, respectively.
- Darbepoetin Alfa: Participants with anemia in CKD who were on hemodialysis received darbepoetin alfa IV once every two weeks up to 26 weeks and received darbepoetin alfa IV twice the dose than earlier, once every month from Week 27 to Week 52.
Period: First Treatment Period
Arm/Group | MIRCERA | Darbepoetin Alfa
Started | 245 | 244
Completed | 216 | 222
Not Completed | 29 | 22
Not completed — Adverse Event | 1 | 2
Not completed — Death | 6 | 7
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Renal transplant | 11 | 7
Not completed — Not defined | 4 | 1
Period: Second Treatment Period
Arm/Group | MIRCERA | Darbepoetin Alfa
Started | 216 | 222
Completed | 187 | 148
Not Completed | 29 | 74
Not completed — Adverse Event | 2 | 5
Not completed — Death | 8 | 4
Not completed — Lack of Efficacy | 9 | 47
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Renal transplant | 4 | 6
Not completed — Not defined | 3 | 8

BASELINE CHARACTERISTICS:
Population: The Safety Population was defined as all participants who received at least one dose of methoxy polyethylene glycol-epoetin beta or darbepoetin alfa and had a safety follow-up, whether withdrawn prematurely or not.
Groups:
- MIRCERA: Participants with anemia in CKD who were on hemodialysis received MIRCERA IV once every month up to 52 weeks. The starting dose of MIRCERA administered during the treatment period was dependent on the dose of darbepoetin alfa administered during screening period and was 120, 200 and 360 mcg/month for weekly darbepoetin alfa doses of <40, 40-80, and >80 mcg, respectively.
- Darbepoetin Alfa: Participants with anemia in CKD who were on hemodialysis received darbepoetin alfa IV once every two weeks up to 26 weeks and received darbepoetin alfa IV twice the dose than earlier, once every month from Week 27 up to Week 52.
- Total: Total of all reporting groups
Arm/Group | MIRCERA | Darbepoetin Alfa | Total
Number analyzed (Participants) | 245 | 244 | 489
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (13.64) | 65.4 (13.91) | 65.8 (13.77)
Gender [Count of Participants; unit: Participants]
  Female | 97 | 89 | 186
  Male | 148 | 155 | 303

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Lesser Than or Equal to One Gram Per Deciliter Decrease in Average Hemoglobin From Baseline and Maintaining Average Hemoglobin Level Greater Than or Equal to 10.5 g/dL Over Evaluation Period
Description: Randomized participants with an average hemoglobin (Hb) decrease from Baseline (Week -4 to Week -1) not exceeding 1.0 gram per deciliter (g/dL) and an absolute average Hb >= 10.5 g/dL during the evaluation period (Weeks 50-53) were defined as responders. Non-responders included participants without any Hb data during the second treatment period and those who did not meet the response criteria and thus were not included in the analysis.
Time Frame: Baseline (Week -4 to Week -1) and Evaluation period (Weeks 50 to 53)
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MIRCERA | Darbepoetin Alfa
Number analyzed (Participants) | 245 | 245
Percentage of participants | 64.1 [57.7 to 70.1] | 40.4 [34.2 to 46.8]
Statistical Analysis 1: Comparison: MIRCERA vs Darbepoetin Alfa; The proportion of responders treated with methoxy polyethylene glycol-epoetin beta versus the proportion of responders treated with darbepoetin alpha during the evaluation period; Test type: Superiority or Other; p < 0.0001, Chi-squared, Corrected; Odds Ratio (OR) = 2.63, 95% CI 2-sided [1.83 to 3.79]

2. Secondary Outcome: Mean Percentage Change in MIRCERA and Darbepoetin Alpha Dose Over Time
Description: All participants received once monthly treatment schedule of both MIRCERA and darbepoetin alpha for the respective treatment arms after Week 27 and these analyses are based on the absolute doses. The average dose in Months 11 and 12 was defined as the mean of all administered doses between study Days 302 and 363. The change in dose was calculated as the percentage change between the respective dose at Week 27 and the average corresponding dose during Months 11 and 12 in each treatment group.
Time Frame: Week 27 to Month 12
Population: ITT population included all randomized participants. Data is presented for the participants available at the time of assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MIRCERA | Darbepoetin Alfa
Number analyzed (Participants) | 211 | 219
percent change | 6.8 (51.0) | 58.8 (76.5)

3. Secondary Outcome: Number of Participants With Marked Laboratory Abnormality Over Time
Description: Values of laboratory parameters higher (H) or lower (L) than the Roche defined reference range were considered as abnormality. The laboratory parameters with abnormality were platelets, white blood cells (WBC), albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), and potassium. Blood samples were drawn before drug administration and before the dialysis session.
Time Frame: Up to Week 53
Population: The Safety Population was defined as all participants who received at least one dose of methoxy polyethylene glycol-epoetin beta or darbepoetin alfa and had a safety follow-up, whether withdrawn prematurely or not. The 'n' represents the number of participants at a specified time point.
Measure: Number; unit: participants
Arm/Group | MIRCERA | Darbepoetin Alfa
Number analyzed (Participants) | 242 | 243
participants
  Platelets-H, n = 241, 243 | 1 | 5
  Platelets-L, n = 241, 243 | 18 | 5
  WBC-H, n = 242, 243 | 4 | 7
  WBC-L, n = 242, 243 | 10 | 4
  ALT-H, n = 241, 242 | 7 | 5
  ALP-H, n = 240, 242 | 12 | 14
  AST-H, n = 239, 240 | 4 | 6
  Albumin-L, n = 240, 242 | 22 | 27
  Phosphate-H, n = 240, 242 | 87 | 92
  Phosphate-L, n = 240, 242 | 36 | 25
  Potassium-H, n = 240, 242 | 54 | 41
  Potassium-L, n = 240, 242 | 2 | 5

4. Secondary Outcome: Median Blood Pressure Over Time
Description: Systolic and diastolic blood pressures (BP) were measured before and after the dialysis session at every week from Baseline (Week -4 to Week -1) to Week 53. Median pre-dialysis diastolic blood pressure (PrD DBP) , median post-dialysis diastolic blood pressure (PoD DBP), median pre-dialysis systolic blood pressure (PrD SBP), and post-dialysis systolic blood pressure (PoD SBP) were reported at Baseline (Week -4 to Week -1) , Week 28 and Week 52.
Time Frame: Baseline (Week -4 to Week -1), Week 28, and Week 52
Population: Safety Population included all participants who received at least one dose of MIRCERA or darbepoetin alfa and had a safety follow-up, whether withdrawn prematurely or not. The 'n' represents the number of participants at a specified time point.
Measure: Median (Full Range); unit: millimeter of mercury
Arm/Group | MIRCERA | Darbepoetin Alfa
Number analyzed (Participants) | 245 | 244
millimeter of mercury
  PrD DBP, Baseline, n = 245, 244 | 75 [32 to 139] | 70 [34 to 206]
  PrD DBP, Week 28, n = 211, 219 | 73 [42 to 118] | 71 [39 to 107]
  PrD DBP, Week 52, n = 187, 147 | 70 [21 to 107] | 70 [39 to 101]
  PoD DBP, Baseline, n = 245, 244 | 70 [33 to 113] | 70 [30 to 132]
  PoD DBP, Week 28, n = 213, 218 | 70 [26 to 101] | 70 [30 to 127]
  PoD DBP, Week 52, n = 186, 148 | 70 [18 to 107] | 65 [33 to 107]
  PrD SBP, Baseline, n = 245, 244 | 140 [83 to 206] | 140 [75 to 241]
  PrD SBP, Week 28, n = 211, 219 | 140 [89 to 219] | 140 [62 to 199]
  PrD SBP, Week 52, n = 187, 147 | 140 [85 to 195] | 132 [84 to 195]
  PoD SBP, Baseline, n = 245, 244 | 133 [83 to 215] | 130 [61 to 248]
  PoD SBP, Week 28, n = 213, 220 | 134 [73 to 228] | 137 [71 to 200]
  PoD SBP, Week 52, n = 186, 148 | 139 [90 to 204] | 127 [70 to 198]

5. Secondary Outcome: Mean Pulse Rate Over Time
Description: Pulse rate is defined as the number of heartbeats in a minute and was assessed in sitting position of the participants at every week from Baseline (Week -4 to Week -1) to Week 53. Summary data of mean values of pulse rate are presented at Baseline (Week -4 to Week -1), Week 28 and Week 52.
Time Frame: Baseline (Week -4 to Week -1), Week 28, and Week 52
Population: The Safety population was defined as all participants who received at least one dose of MIRCERA or darbepoetin alfa and had a safety follow-up, whether withdrawn prematurely or not. The 'n' represents the number of participants at a specified time point.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | MIRCERA | Darbepoetin Alfa
Number analyzed (Participants) | 245 | 244
beats per minute
  Baseline, n = 245, 244 | 73 (11.1) | 73 (12.3)
  Week 28, n = 211, 215 | 74 (13.0) | 72 (12.6)
  Week 52, n = 184, 147 | 73 (12.5) | 71 (11.3)

6. Secondary Outcome: Number of Participants With Any Adverse Events, Serious Adverse Events, and Deaths
Description: An adverse event (AE) can be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. A serious adverse event (SAE) is any adverse event that can result in death or is life-threatening or required in participants hospitalization or prolongation of existing hospitalization or results in persistent or significant disability/incapacity; or is a congenital anomaly/birth defect; or is medically significant or requires intervention to prevent one or other of the outcomes listed above. SAEs were reported up to Week 56, while nonserious AEs up to Week 52.
Time Frame: From screening to Week 56
Population: The Safety Population was defined as all participants who received at least one dose of MIRCERA or darbepoetin alfa and had a safety follow-up, whether withdrawn prematurely or not. Among the 14 deaths in Darbepoetin alfa group, 3 participants died after withdrawal from the study and within 30 days after last dose of study drug.
Measure: Number; unit: Participants
Arm/Group | MIRCERA | Darbepoetin Alfa
Number analyzed (Participants) | 245 | 244
Participants
  Participants with any AE | 222 | 217
  Participants with any SAE | 99 | 94
  Deaths | 14 | 14

ADVERSE EVENTS:
Time Frame: Up to Week 56
Description: The Safety Population was defined as all participants who received at least one dose of methoxy polyethylene glycol-epoetin beta or darbepoetin alfa and had a safety follow-up, whether withdrawn prematurely or not. SAEs were reported up to Week 56; however, nonserious AEs were reported up to Week 52 only.
Arm/Group | MIRCERA | Darbepoetin Alfa
Serious Adverse Events (participants affected / at risk) | 99/245 | 94/244
Other Adverse Events (participants affected / at risk) | 140/245 | 126/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MIRCERA (N=245) | Darbepoetin Alfa (N=244)
Sepsis (Infections and infestations) | 3 | 5
Pneumonia (Infections and infestations) | 3 | 4
Bronchitis (Infections and infestations) | 3 | 1
Gastroenteritis (Infections and infestations) | 2 | 2
Catheter related infection (Infections and infestations) | 1 | 2
Catheter sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 2 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Abscess limb (Infections and infestations) | 0 | 1
Arteriovenous graft site infection (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Central line infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Implant site abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Post procedural sepsis (Infections and infestations) | 1 | 0
Post operative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Arteriovenous Fistula site complication (Injury, poisoning and procedural complications) | 8 | 5
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 10 | 2
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 | 4
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 | 2
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 2
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Procedural Hypotension (Injury, poisoning and procedural complications) | 1 | 1
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Stent occlusion (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Myocardial infarction (Cardiac disorders) | 4 | 3
Acute coronary syndrome (Cardiac disorders) | 2 | 3
Atrial fibrillation (Cardiac disorders) | 3 | 2
Angina pectoris (Cardiac disorders) | 2 | 2
Angina unstable (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Electromechanical dissociation (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Postinfarction angina (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 3 | 2
Arterial occlusive disease (Vascular disorders) | 0 | 4
Hypertensive crisis (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Arteriosclerosis obliterans (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Diabetic vascular disorder (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Microscopic polyangiitis (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Faecalith (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal telangiectasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 3
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Vascular dementia (Nervous system disorders) | 0 | 2
Basilar artery thrombosis (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Ischaemic neuropathy (Nervous system disorders) | 0 | 1
Myxoedema coma (Nervous system disorders) | 1 | 0
Neurodegenerative disorder (Nervous system disorders) | 1 | 0
Periodic limb movement disorder (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Uraemic encephalopathy (Nervous system disorders) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meigs' syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neurilemmoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 1
Fluid overload (Metabolism and nutrition disorders) | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Catheter thrombosis (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Multi-Organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 3
Renal haemorrhage (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 2
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Hyperparathyroidism Secondary (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Amyloidosis (Immune system disorders) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MIRCERA (N=245) | Darbepoetin Alfa (N=244)
Nasopharyngitis (Infections and infestations) | 25 | 20
Urinary tract infection (Infections and infestations) | 23 | 15
Bronchitis (Infections and infestations) | 17 | 16
Influenza (Infections and infestations) | 13 | 17
Procedural hypotension (Injury, poisoning and procedural complications) | 20 | 26
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 16 | 15
Diarrhoea (Gastrointestinal disorders) | 17 | 19
Nausea (Gastrointestinal disorders) | 14 | 8
Constipation (Gastrointestinal disorders) | 16 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 13
Hypertension (Vascular disorders) | 35 | 26
Fluid overload (Metabolism and nutrition disorders) | 9 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.